CLINICAL TRIAL: NCT07340723
Title: Novel First-line Therapies for Grade II Acute GVHD: a Randomized Controlled Trial
Brief Title: Novel First-line Therapies for Grade II Acute GVHD(Graft-versus-host Disease )
Acronym: GVHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daihong Liu (Other)
Responsible Party: Sponsor-Investigator, Daihong Liu, Department of Hematology, Senior Department of Hematology, The Fifth Medical Center of PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2025-767-01
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-06

CONDITIONS: GVHD,Acute; Stem Cell Transplant Complications
Keywords: acute graft-versus-host disease; Ruxolitinib; first line therapy
MeSH Terms: interventions — ruxolitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Drug:Ruxolitinib, Corticosteroids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib Arm (Experimental): Ruxolitinib combined with Corticosteroids
  Interventions: Drug: Ruxolitinib; Drug: Corticosteroids
- Comparator arm (Active Comparator)
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Drug: Ruxolitinib — Participants began oral administration of ruxolitinib at 5 mg QD;Methylprednisolone: 0.5mg/kg/d , iv or iv gtt for at least 5 days, then taper according to the clinical response.
  Arms: Ruxolitinib Arm
Drug: Corticosteroids — Methylprednisolone: 2mg/kg/d , iv or iv gtt for at least 1 week, then taper according to the clinical response.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of combined Ruxolitinib With Corticosteroids as First Line Therapy for grade II acute GVHD (graft-versus-host disease )

DETAILED DESCRIPTION:
Acute graft-versus-host disease (GVHD) is treated with systemic corticosteroid immunosuppression as first line therapy. Many patients with grade II acute GVHD do not respond to primary therapy, high-dose systemic corticosteroids; therefore, survival for those patients remains particularly poor. Here we determine the efficacy and safety of combined Ruxolitinib With Corticosteroids as First Line Therapy for the Treatment of grade II acute GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hematological diseases.
2. Have undergone first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies.
3. New onset of grade II acute GVHD or intermediate or high risk aGVHD (based on modified GVHD Glucksberg criteria) within 100 days post-transplantation.

Exclusion Criteria:

1. Recipients of second allogeneic stem cell transplant.
2. Acute GVHD induced by donor lymphocyte infusion, interferon.
3. Received first line aGVHD treatment before enrollment.
4. Overlap GVHD syndrome.
5. Pregnant or breast-feeding women.
6. Pregnant or breast-feeding women.
7. Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockroft-Gault equation.
8. Uncontrolled infection.
9. Human immunodeficiency virus infection.
10. Active hepatitis b virus, hepatitis C virus infection and need antivirus treatment.
11. Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed, or graft rejection.
12. Allergic history to Janus kinase inhibitors.
13. Severe organ dysfunction unrelated to underlying GVHD, including:

(1)Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction).

(2)Clinically significant or uncontrolled cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy.

(3)Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.

14.Received Janus kinase inhibitor therapy after allo-HSCT for any indication. 15.Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) at Day 28 | Day 28 after treatment
  Defined as the proportion of participants demonstrating a complete response (CR), or partial response (PR).

SECONDARY OUTCOMES:
Six-month duration of response | Six-month after treatment
  Defined as the time from first response until graft-versus-host disease (GVHD) progression or death. Six-month duration of response will be assessed when all participants who are still on study complete the Day 180 visit.
Duration of response | Day 90 after treatment
  Defined as the time from first response until GVHD progression or death, when all participants who are still on study complete the Day 90 visit.
Nonrelapse mortality (NRM) | 1 year after treatment
  NRM was deﬁned as death from any cause without relapse. Cumulative incidence of NRM was analyzed in a competing risk framework using Gray's method.
Cumulative incidence of relapse (CIR) | 1 year after treatment
  Defined as the proportion of participants whose underlying malignancy relapsed.Relapse was defined as hematologic recurrence of malignancies after transplantation. Cumulative incidence of relapse was analyzed in a competing risk framework using Gray's method.
Disease-free survival (DFS) | 1 year after treatment
  Defined as the time from day +1 to the earliest date that a participant died, had a relapse/progression of the underlying malignancy, required additional therapy for aGVHD, or demonstrated signs or symptoms of chronic graft-versus-host disease (cGVHD).DFS will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test.
Overall survival (OS) | 1 year after treatment
  Defined as survival from day +1 until death or last follow-up. OS will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test. Survival will be calculated from the date of randomization.
GVHD-free and relapse-free survival (GRFS) | 1 year after treatment
  Defined as a composite endpoint of death from any cause, disease relapse, grade Ⅲ-Ⅳ acute GVHD, or chronic GVHD requiring systemic immunosuppression therapy.
Recurrence of aGVHD | 1 year after treatment
  Defined as the proportion of participants whose aGVHD relapsed.Relapse was defined as recurrence of new GVHD related symptoms after complete remission of aGVHD. Cumulative incidence of recurrence of aGVHD was analyzed in a competing risk framework using Gray's method.
Failure-free survival | 1 year after treatment
  Failure-free survival (FFS) refers to the time from day +1 to disease relapse or progression, non-relapse mortality, or the addition of new therapy for aGVHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Senior Department of Hematology, The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data requests should be evaluated on a case-by-case basis by an independent review committee in accordance with the moderated access policy of the Data Repository Unit at the Chinese PLA General Hospital, Beijing, China.

REFERENCES:
- [Background] von Bubnoff N, Ihorst G, Grishina O, Rothling N, Bertz H, Duyster J, Finke J, Zeiser R. Ruxolitinib in GvHD (RIG) study: a multicenter, randomized phase 2 trial to determine the response rate of Ruxolitinib and best available treatment (BAT) versus BAT in steroid-refractory acute graft-versus-host disease (aGvHD) (NCT02396628). BMC Cancer. 2018 Nov 19;18(1):1132. doi: 10.1186/s12885-018-5045-7. PMID 30453910
- [Background] Zeiser R, von Bubnoff N, Butler J, Mohty M, Niederwieser D, Or R, Szer J, Wagner EM, Zuckerman T, Mahuzier B, Xu J, Wilke C, Gandhi KK, Socie G; REACH2 Trial Group. Ruxolitinib for Glucocorticoid-Refractory Acute Graft-versus-Host Disease. N Engl J Med. 2020 May 7;382(19):1800-1810. doi: 10.1056/NEJMoa1917635. Epub 2020 Apr 22. PMID 32320566
- [Background] Kujawska J, Zeiser R, Gil L. Recent advances in acute gastrointestinal graft versus host disease (aGvHD): aspects of steroid-resistant disease. Ann Hematol. 2025 Feb;104(2):855-865. doi: 10.1007/s00277-024-05952-0. Epub 2024 Aug 29. PMID 39207560
- [Background] Holtan SG, Yu J, Choe HK, Paranagama D, Tang J, Naim A, Galvin J, Joachim Deeg H. Disease progression, treatments, hospitalization, and clinical outcomes in acute GVHD: a multicenter chart review. Bone Marrow Transplant. 2022 Oct;57(10):1581-1585. doi: 10.1038/s41409-022-01764-w. Epub 2022 Jul 30. PMID 35908108
- [Background] Dou L, Zhao Y, Yang J, Deng L, Wang N, Zhang X, Liu Q, Yang Y, Wei Z, Wang F, Jiao Y, Li F, Luan S, Hu L, Gao S, Liu C, Liu X, Yan J, Zhang X, Zhou F, Lu P, Liu D. Ruxolitinib plus steroids for acute graft versus host disease: a multicenter, randomized, phase 3 trial. Signal Transduct Target Ther. 2024 Oct 23;9(1):288. doi: 10.1038/s41392-024-01987-x. PMID 39438467